CLINICAL TRIAL: NCT03697512
Title: MALIBU Trial - Phase II Study of Combination Ibrutinib and Rituximab in Untreated Marginal Zone Lymphomas
Brief Title: MALIBU Trial - Combination of Ibrutinib and Rituximab in Untreated Marginal Zone Lymphomas
Acronym: MALIBU
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG47; 2018-002364-44 (EudraCT Number)
Record Dates: First submitted 2018-09-28; First posted 2018-10-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Marginal Zone Lymphoma; Nodal Marginal Zone Lymphoma; Splenic Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — ibrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ibrutinib and Rituximab (Experimental): Induction PART A, from Day 1 to Day 56.
  Patients will be treated with:
  * Ibrutinib 560 mg/day continuously up to Day 56;
  * Rituximab 375 mg/m2 intravenously at Day 1, and then subcutaneous (1400 mg, flat dose) at Day 8, 15 and 22 of cycle 1.
  Induction PART B, from Day 57 to Day 196.
  Patients will be treated with:
  * Ibrutinib 560 mg/day continuously up to Day 196;
  * Rituximab subcutaneous (1400 mg, flat dose) at Day 1 every 28 days for 4 cycles.
  Maintenance PART C, from Day 197 to Day 730.
  Patients will be treated with:
  - Ibrutinib 560 mg/day continuously up to Day 730.
  Interventions: Drug: Ibrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — capsules for oral intake in a dosage of 560 mg (four capsules) daily
Drug: Rituximab — Concentrate solution for infusion - intravenous use; Solution for injection - subcutaneous use.

SUMMARY:
Single-arm, phase II clinical trial of patients with Extranodal Marginal Zone Lymphoma (EMZL). It is planned to recruit 130 patients.

Additional patients with Splenic Marginal Zone Lymphoma (SMZL), up to 30, and Nodal Marginal Zone Lymphoma (NMZL), up to 15, will be included in the trial in order to preliminary explore the clinical activity and safety of the combination treatment proposed.

The study primary endpoints will be analysed on the EMZL population. Outcome of patients with SMZL and NMZL will be analysed and reported separately

DETAILED DESCRIPTION:
Marginal zone lymphomas (MZL) represent a group of indolent B-cell lymphomas that arises from marginal zone B-cells in extranodal tissues, such as spleen and mucosa associated lymphoid tissues, and more rarely also in nodal tissues. MZL comprises 5 to 17% of all non-Hodgkin lymphomas (NHL) in adults. The 2016 World Health Organization (WHO) recognized three separate subtypes of MZL according to their primary localization, namely the:

1. extranodal MZL (EMZL) of mucosa-associated lymphoid tissue (MALT), also known as MALT lymphoma
2. splenic MZL (SMZL)
3. nodal MZL (NMZL). These three subtypes are distinct disease entities that are classified together because they all seem to originate from post germinal centre marginal zone B-cells.

MALIBU trial is a prospective multicenter trial combining rituximab and ibrutinib in front-line for patients with MZL, including EMZL, SMZL and NMZL Aim of the study is to assess the safety and efficacy of the combination of rituximab and ibrutinib in EMZL patients and to explore its activity in SMZL and NMZL as exploratory subset.

ELIGIBILITY:
Inclusion Criteria:

Chemotherapy and immunotherapy-naïve, symptomatic and in need of treatment patients, with histologically proven CD20-positive MZL, not eligible for local therapy, including:

1. EMZL (MALT Lymphoma) patients with MALT- IPI score 1-2 in need of systemic therapy.

   Either de novo or relapsed following local therapy (including surgery, radiotherapy and antibiotics for H. pylori-positive gastric lymphoma) arisen at any extranodal site with MALT-international prognostic index (IPI) score 1-2 at the time of study entry.

   1.1.The following patients with gastric MALT Lymphoma can be entered:
   1. H. pylori-negative cases, either de novo (non pretreated) or at relapse following local therapy (i.e., surgery, radiotherapy or antibiotics).
   2. H. pylori-positive cases at diagnosis, who either first line antibiotics or further local treatment (surgery or radiotherapy), including patients with:

      * clinical (endoscopic) and histological evidence of disease progression at any time post H. pylori eradication;
      * clinical (endoscopic) and histological relapse (without H. pylori re-infection), after a remission patients;
      * persistent (stable) lymphoma at ≥ 1 year post H. pylori eradication. 1.2. Similar consideration may be applied to patients with ocular adnexal lymphoma treated with antibiotics.
2. SMZL patients in need of therapy. Either de novo or relapsed following local therapy [including surgery and antiviral therapy for Hepatitis C virus (HCV)]. Patient must have a symptomatic disease requiring treatment and be not eligible for splenectomy or not willing to undergo splenectomy.

   2.1. Patients with SMZL can be entered if any of the following criteria is present:
   1. bulky progressive or painful splenomegaly;
   2. enlarged lymph nodes or involvement of extranodal sites with or without cytopenias , i.e. involvement of ≥3 nodal sites, each with a diameter of ≥3 cm. Any nodal tumor mass with a diameter of ≥7 cm (GELG criteria, as adopted in follicular lymphoma);
   3. one of the following symptomatic/progressive cytopenias:

      * Hgb < 10 g/dL;
      * ANC < 1000/μL:
      * PLT< 80 000/μL whatever the reason (autoimmune or hypersplenism or bone marrow infiltration).

   2.2. Splenectomised patients with rapidly raising lymphocyte counts, lymphadenopathy or involvement of extranodal sites can be entered.

   2.3. SMZL with concomitant HCV infection who have not responded to or are relapsed after antiviral therapy can be entered.
3. NMZL patients in need of therapy Either, de novo presenting with disseminated disease or relapsed after local radiotherapy or following antiviral therapy for HCV. Localized nodal MZL is not eligible.

   * Measurable or evaluable disease.
   * Ann Arbor II-IV. Stage I disease may be eligible only if not candidate to local therapy (surgery or radiotherapy).
   * Age ≥ 18.
   * Life expectancy of at least 1 year.
   * ECOG Performance status 0-2.
   * Adequate bone marrow, kidney and liver function
   * For women of childbearing potential only: negative serum pregnancy test done within 7 days prior to study drugs administration or within 14 days if with a confirmatory urine pregnancy test within 7 days prior to the first study drugs administration.
   * Fertile male or female patients of childbearing potential and their partners must use higly effective contraception methods during the study and for at least 12 months after the last dose of subcutaneous rituximab. In case hormonal methods of birth control is used a barrier method must be added.
   * Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Any type of lymphoma other than MZL (including MZL with histologic transformation to high-grade lymphoma).
2. Localized (stage IE and IIE) MALT lymphoma, for example gastric, ocular and cutaneous lymphoma, that may benefit from local therapy only (surgery or radiotherapy).
3. Known CNS involvement of MZL.
4. Any previous systemic treatment with immunotherapy or chemotherapy or with BTK inhibitors.
5. Major surgery within 4 weeks prior to registration.
6. History of stroke or intracranial bleeding within 6 months.
7. Known bleeding diathesis (eg, von Willebrand's disease) or hemophilia.
8. Concurrent use of warfarin of other vitamin K antagonists.
9. Concurrent use of strong cytochrome P450 (CYP)3A4/5 inhibitors (see http://medicine.iupui.edu/clinpharm/ddis/clinical-table/).
10. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.
11. International normalized ratio (INR) or prothrombin time (PT) ≥1.5 ULN. Partial thromboplastin time (PTT) or activated PTT (aPTT) ≥1.5 ULN unless due to lupus anticoagulant.
12. Vaccinated with live, attenuated vaccines within 4 weeks prior to randomization.
13. Clinically significant hypersensitivity (e.g., anaphylactic or anaphylactoid reactions to the compound of ibrutinib and/or rituximab themselves or to the excipients in their formulation).
14. Positive test results for chronic HBV infection (defined as positive HBsAg serology).
15. Patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) may be included if HBV DNA is undetectable, provided that they are willing to undergo monthly DNA testing and taking specific antiviral prophylaxis, according to local policy. Patients who have protective titers of hepatitis B surface antibody (HBsAb) after vaccination are eligible.
16. Positive test results for hepatitis C. Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
17. HIV infection or immunodeficiency.
18. Active, severe infections
19. Pregnancy or breastfeeding.
20. Clinically significant cardiovascular diseases such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
21. Any serious medical or psychiatric illness likely to interfere with participation in this clinical study.
22. Prior history of malignancies other than MZL within 3 years,with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer.
23. Current enrolment or participation in another therapeutic clinical trial within 28 days prior to treatment start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate at 12 months | 12 months after treatment start
  The proportion of patients with complete response after 12 months from treatment start
Progression Free Survival at 5 years | 5 years from treatment start
  The proportion of patients without disease progression after 5 years from treatment start

SECONDARY OUTCOMES:
Number of treatment-Emerging Adverse Events | From the time of informed consent signature until 28 days after treatment discontinuation or until resolution of all treatment-related AEs, whichever occurs later
  Analysis of incidence, severity and relationship of adverse events graded according to NCI Common Toxicity Criteria, version 4.0
Complete Response Rate at 24 months | 24 months from treatment start
  The proportion of patients with complete response after 24 months from treatment start
Overall Response Rate at 12 and 24 months | 12 and 24 months after treatment start
  The proportion of responding patients (partial and complete responses) assessed at 12 and 24 months after treatment start
Overall survival | From the date of treatment start to the date of death due to any cause until 5 years from treatment discontinuation
  The time from the date of treatment start to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Thieblemont, MD, Study Chair — Saint-Louis Hospital, Paris, France; Annarita Conconi, MD, Study Chair — Ospedale degli Infermi - Biella, Italy
Locations (36):
- CHU UCL Namur / site Godinne, Yvoir, Belgium
- France (13):
  - CHU de Tours - Hôpital Bretonneau, Tours, Cedex 01
  - CHU de Montpellier, Montpellier, Cedex 05
  - CHU d'Estaing, Clermont-Ferrand, Cedex 1
  - CHU de Rennes Pontchaillou, Rennes, Cedex 9
  - Institut Bergonié, Bordeaux
  - IHBN - CHU Côte de Nacre, Caen
  - CHU Dijon Bourgogne - Hôpital François Mitterand, Dijon
  - CHU de Grenoble - Hôpital Albert MICHALLON, La Tronche
  - Saint Louis Hospital, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHRU de Strasbourg, Strasbourg
  - IUCT Oncopole Toulouse, Toulouse
  - CHU de Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy
- Italy (16):
  - Ospedale degli Infermi, Ponderano, BI
  - Ospedale San Raffaele, Milan, MI
  - A.O.U. Città della Salute e della Scienza di Torino Ospedale Molinette, Torino, TO
  - Azienda Ospedaliera Universitaria Ospedali Riuniti - Università Politecnica delle Marche, Ancona
  - Giovanni Paolo II/I.R.C.C.S. Istituto Tumori, Bari
  - A.O. Spedali Civili di Brescia, Brescia
  - Ospedale Oncologico Businco, Cagliari
  - Fondazione IRCCS - Cà Granda - Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - AAST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS - Policlinico San Matteo, Pavia
  - U.O. Ematologia AUSL Ravenna, Ravenna
  - Azienda Ospedaliera Arcispedale Santa Maria Nuova IRCCS, Reggio Emilia
  - Università degli Studi di Roma La Sapienza, Roma
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI), Trieste
  - Ospedale di Circolo e Fondazione Macchi di Varese, Varese
- Instituto Português de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon, Portugal
- Switzerland (5):
  - Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona, Canton Ticino
  - Kantonalspital Baden, Baden
  - Inselspital Bern, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - Universitätsspital Zürich, Zurich